CLINICAL TRIAL: NCT00212316
Title: Phenylbutyrate Development for Huntington's Disease (PHEND-HD): A Multi-Center, Double-Blind, Placebo-Controlled Study With Open-Label Follow-Up to Determine the Safety and Tolerability of Phenylbutyrate in Subjects With Huntington's Disease
Brief Title: Safety and Tolerability Study of Phenylbutyrate in Huntington's Disease (PHEND-HD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: HP Therapeutics Foundation (Other); Massachusetts General Hospital (Other); Columbia University (Other); University of Iowa (Other); University of California, San Diego (Other); University of Kansas (Other); University of Alabama at Birmingham (Other); Johns Hopkins University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01NS45242
Record Dates: First submitted 2005-09-19; First posted 2005-09-21 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2007-12

CONDITIONS: Huntington's Disease
Keywords: Huntington's Disease; phenylbutyrate; HDAC inhibitors; transcription
MeSH Terms: conditions — Huntington Disease | interventions — 4-phenylbutyric acid

INTERVENTIONS:
Drug: sodium phenylbutyrate

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and clinical impact of 15-grams daily of sodium phenylbutyrate (phenylbutyrate) in Huntington's disease and to lay the groundwork for possible subsequent trials designed to specifically address its ability to slow or halt the progression of the disease.

DETAILED DESCRIPTION:
Huntington's disease (HD) is an autosomal dominant disorder resulting in selective loss of neurons in the striatum-an area of the brain that controls movement, balance, and walking-and other areas of the brain. The disease is characterized by progressive motor and cognitive decline. There is no cure or even plausible treatment to offset the fatal course of the disease. Therefore, any treatment that ameliorates the disease would be of enormous importance.

The purpose of this double-blind, placebo-controlled study-with open-label follow-up-is to determine the safety and tolerability of 15-grams daily of oral phenylbutyrate in people with HD. The study will enroll 60 individuals. Eligible participants will be initially randomized to receive either phenylbutyrate or the matching placebo for 4 weeks.

After the placebo-controlled phase, all participants will enter the open-label phase to receive phenylbutyrate for 12 weeks. Participants will be followed for one month off phenylbutyrate.

This combination of a short-term double-blind, placebo-controlled phase followed by a longer open-label phase will favor the primary goals of detecting toxicity and intolerability while facilitating recruitment and maximizing number of subjects on study drug.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with clinical diagnosis of HD and family history of HD or a CAG repeat expansion greater than or equal to 37
* Subjects in stage I or II of illness (TFC greater than or equal to 7)
* Subjects must be ambulatory and not requiring skilled nursing care
* Age of 18 years or older
* Women of childbearing potential (i.e., those not postmenopausal or surgically sterile) must confirm to the best of their knowledge that they are not pregnant or plan to get pregnant
* Women of childbearing potential must have negative pregnancy test, be non-lactating and use adequate contraception methods, such as oral birth control pills plus a barrier method (i.e. condoms, diaphragm) or IUD during their participation in the study
* Subjects currently taking psychotropic medications (including antidepressants and neuroleptics) must be on stable dosages for at least 4 weeks prior to baseline visit and should be maintained on constant dosage throughout the study
* Subjects must be capable of providing informed consent and complying with trial procedures
* Subjects must be able to take oral medication, a person willing and able to serve as an informant and provide information about the daily dosing of study medication

Exclusion Criteria:

* Exposure to phenylbutyrate, valproic acid, probenecid, known HDAC inhibitors or other transcriptionally active compounds within 3 months (90 days) prior to the baseline visit
* History of known sensitivity or intolerability to phenylbutyrate, sodium butyrate or sodium acetate
* Existence of a known malignancy that might require treatment during the course of this study
* Exposure to any investigational drug within 30 days of the baseline visit
* Subjects with underlying hematologic, hepatic or renal disease; screening white blood cell (WBC) count less than 3,800/mm3, screening creatinine greater than 2.0 or alanine aminotransferase (ALT) greater than 2 times the upper limit of normal
* Clinical evidence of unstable medical illness in the investigator's judgment
* Clinical illness that requires use of warfarin (Coumadin)
* Unstable psychiatric illness defined as psychosis (hallucinations or delusions) untreated major depression or plan for suicide within 90 days of the baseline visit
* Current or history of substance (alcohol or drug) abuse within 1 year of the baseline visit
* Pregnant women or women who are currently breast-feeding
* History of heart failure or other conditions that might be exacerbated by sodium loading

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-08; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects able to complete treatment (Week 16)

SECONDARY OUTCOMES:
Secondary safety and tolerability outcomes at Weeks 1, 4, 5, 10, 16, & 20 include:
adverse events,
changes in vital signs,
and clinical lab assessments.
Secondary clinical measures at Weeks 4, 10, 16, and 20 include components of the UHDRS:
total motor,
Stroop,
independence,
& total functional capacity.
Secondary biological indicators of treatment affects at Weeks 4, 10, 16, & 20 include:
markers of neuroprotection (e.g. NAA) via MRS,
histone acetylation (levels in WBC; fetal hemoglobin levels in blood),
depletion of glutamine,
gene expression analyses,
and biochemical analyses for pharmacokinetics.

CONTACTS AND LOCATIONS:
Overall Officials: Steven M. Hersch, MD, PhD, Principal Investigator — Co-Chair, Huntington Study Group, Massachusetts General Hospital; Karl Kieburtz, MD, MPH, Principal Investigator — Director, Clinical Trials Coordination Center, University of Rochester
Locations (8):
- United States (8):
  - University of Alabama, Birmingham, Alabama
  - University of California-San Diego, San Diego, California
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Columbia University, New York, New York
  - University of Rochester, Rochester, New York